CLINICAL TRIAL: NCT01367184
Title: IVC Filter Study to Monitor and Measure Patients Outcomes Through Standardized Collection and Analysis of Clinical Information
Brief Title: National Inferior Vena Cava (IVC) Filter Registry
Status: Terminated | Type: Observational
Sponsor: American Venous Forum (Other)
Responsible Party: Sponsor
Other Study IDs: AVR-IVC-01
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Venous Thrombo-embolism
Keywords: VTE; Inferior vena cava; Venous thrombo-embolism; Outcome data; IVC Filters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Inferior vena cava (IVC) filter is an important therapeutic device used in the management of venous thrombo-embolism (VTE) in patients that are contra-indicated for anti-coagulation therapy. While there has been significant increase in the use of filters , unfortunately there are no standardized collection of data to track, compare outcomes, report safety and efficacy.

DETAILED DESCRIPTION:
The registry is a multi-institutional bioinformatics database for the collection of data relevant to Inferior vena cava filters. Participating study centers may enroll patients and enter data in the web-based registry that include demographics, clinical features, management details and follow-up up to 48 months.

The purpose of this study is to improve our understanding of the retrieval rate, long term safety and efficacy on IVC filters placed in North America.

ELIGIBILITY:
Inclusion Criteria:

* Data obtained in line with good clinical practice,applicable laws and regulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No specific criteria. Data from anyone who underwent IVC Filter Placement/Retrieval will be eligible
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Integrity of IVC Filter 12 months post placement | 48 Months

CONTACTS AND LOCATIONS:
Overall Officials: Brajesh K Lal, Study Chair — University of Maryland Medical Center,Baltimore; John E. Rectenwald, Principal Investigator — University of Michigan; Uchenna N Onyeachom, Study Director — American Venous Forum
Locations (27):
- United States (27):
  - Exempla Lutheran Medical Center, Denver, Colorado
  - University of Florida , Division of Vascular Surgery & Endovascular Therapy, Gainesville, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - Medical Center of Central Georgia, Macon, Georgia
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - University of Chicago Hospitals, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University Of Kentucky , Vascular and Endovascular Divison, Lexington, Kentucky
  - Tuoro Infirmary, New Orleans, Louisiana
  - University Of Michigan Health System, Ann Arbor, Michigan
  - St. Luke's Medical Center, Chesterfield, Missouri
  - St Peters Hospital, Helena, Montana
  - Brooklyn Hospital, New York, New York
  - University Of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Vein Clinic, Stony Brook, New York
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pittsburgh School of Medicine Division of Vascular Surgery, Pittsburgh, Pennsylvania
  - Palmetto Health and Providence Hospital, Columbia, South Carolina
  - Vascular Health Alliance, Greenville Hospital System, Greenville, South Carolina
  - Avera Sacred Heart Hospital, Yankton, South Dakota
  - Northwest Texas Hospital, Amarillo, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Intermountain Medical Center, Murray, Utah
  - West Virginia University Healthcare, Morgantown, West Virginia

REFERENCES:
- See also: Related Info — http://www.venousregistry.org